CLINICAL TRIAL: NCT04318782
Title: A Prospective Study for the Treatment of Severe Pulmonary Embolism With Pharmacodynamic Thrombectomy
Acronym: RESPIRE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P171007J; 2019-A01627-50 (Other: ANSM); DR-2019-329 (Other: CNIL)
Record Dates: First submitted 2020-03-20; First posted 2020-03-24 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Pulmonary Embolism
Keywords: pulmonary embolism; pharmacodynamic thrombectomy; endovascular embolectomy
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Thrombectomy (Experimental): Pharmacodynamic thrombectomy using AngioJet ™ PE Thrombectomy Catheter
  Interventions: Device: Pharmacodynamic thrombectomy

INTERVENTIONS:
Device: Pharmacodynamic thrombectomy — Pharmacodynamic thrombectomy using AngioJet ™ PE Thrombectomy Catheter

SUMMARY:
The mortality of severe pulmonary embolisms admitted to the resuscitation department for circulatory failure remains in the range of 30-40% at the acute phase. Hemodynamic failure is the leading cause of death. These patients frequently have a contraindication to thrombolysis. Surgical pulmonary arterial desobstruction still leads to significant hospital mortality and can't be implemented in all hospitals. Concerning advanced hemodynamic support techniques, they can't always reduce mortality on themselves. There is therefore a need for developing alternative approaches for less invasive pulmonary arterial desobstruction. Data on the efficacy and safety of percutaneous methods of desobstruction are still too limited to implement them in current practice.

AngioJet ™ PE is a device CE marked for intra-arterial desobstruction of pulmonary arteries. It has been successfully tested in more than 25 patients with pulmonary embolism in France. Before considering a request for reimbursement from the HAS it is necessary to have propective data of sufficient quality. This phase 2a prospective study is proposed to evaluate the efficacy and safety of the AngioJet ™ PE catheter use. The resulting data will allow us to submit a Phase 3 controlled study to an upcoming PHRC-type project call.

ELIGIBILITY:
Inclusion Criteria:

* Pulmonary embolism objectively confirmed by thoracic angioTDM
* Date of onset of pulmonary embolism 14 days prior to inclusion
* State of shock
* Presence of at least 6 mm thrombus in a main or lobar pulmonary artery
* Contraindication (absolute or relative) or systemic fibrinolysis treatment failure defined by persistence of shock, as defined above, more than 6 hours

Exclusion Criteria:

* Known cardiac pathologies with right-left cardiac shunt
* Target pulmonary artery 6 mm in diameter
* Known heparin allergy or thrombocytopenia
* Known severe hypersensitivity to iodine contrast products
* Severe renal failure defined by creatinine clearance 30 ml/min Pregnant or lactating patient
* Patient not affiliated to social security
* Patient with unhealed lesion due to recent mechanical intervention on the vessel to be treated

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-02-10 (Actual); Primary Completion 2021-02-10 (Estimated); Study Completion 2021-02-10 (Estimated)

PRIMARY OUTCOMES:
Survival rate | one month
  Survival rate at one month

SECONDARY OUTCOMES:
Global mortality | 7 days
  Global mortality at 7 days
Global mortality | 30 days
  Global mortality at 30 days
Pulmonary Embolism mortality | 7 days
  Pulmonary Embolism mortality at 7 days
Pulmonary Embolism mortality | 30 days
  Pulmonary Embolism mortality at 30 days
Major bleeding rate | 7 days
  Major bleeding rate at 7 days
Major bleeding rate | 30 days
  Major bleeding rate at 30 days
Clinically significant non-major bleeding | 7 days
  Clinically significant non-major bleeding at 7 days
Clinically significant non-major bleeding | 30 days
  Clinically significant non-major bleeding at 30 days
Thromboembolic recurrence rate | 7 days
  Objectively confirmed thromboembolic recurrence rate at 7 days
Thromboembolic recurrence rate | 30 days
  Objectively confirmed thromboembolic recurrence rate at 30 days
Cumulative rate of patients requiring a surgical pulmonary thrombectomy | 7 days
  Cumulative rate of patients requiring a surgical pulmonary thrombectomy at 7 days
Cumulative rate of patients requiring a surgical pulmonary thrombectomy | 30 days
  Cumulative rate of patients requiring a surgical pulmonary thrombectomy at 30 days
Clinical success rate | 7 days
  Clinical success rate at 7 days
Clinical success rate | 30 days
  Clinical success rate at 30 days
Description of AE/SAE | 30 days
  Description of AE/SAE at 30 days
Modification of the ratio of right/left ventricle diameter | 48 hours
  Modification of the ratio of right/left ventricle diameter at 48 hours
Modification of the scanographic pulmonary vascular obstruction score | 48 hours
  Modification of the scanographic pulmonary vascular obstruction score at 48 hours
Results of coagulation / fibrinolysis markers | 7 days
  Results of coagulation / fibrinolysis markers at 7 days
Results of coagulation / fibrinolysis markers | 30 days
  Results of coagulation / fibrinolysis markers at 30 days
Length of hospital stay | 30 days
  Length of hospital stay
Length of stay in the intensive care unit | 30 days
  Length of stay in the intensive care unit

CONTACTS AND LOCATIONS:
Overall Officials: DEL GIUDICE Costantino, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- AP-HP - Hôpital Européen Georges-Pompidou Paris, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in publication could be shared Individual participant data detailed in meta analysis protocol could be shared
Supporting Information: Study Protocol, ICF
Time Frame: One year after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on scientific project and scientific involvement of the PI team.
  Teams wishing obtain IPD must meet the sponsor and IP team to present scientifics (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractualization